CLINICAL TRIAL: NCT03371381
Title: An Open-Label Randomized Phase 1b/2 Study of the Efficacy and Safety of JNJ-64041757, a Live Attenuated Listeria Monocytogenes Immunotherapy, in Combination With Nivolumab Versus Nivolumab Monotherapy in Subjects With Advanced Adenocarcinoma of the Lung
Brief Title: An Efficacy and Safety Study of JNJ-64041757, a Live Attenuated Listeria Monocytogenes Immunotherapy, in Combination With Nivolumab Versus Nivolumab Monotherapy in Participants With Advanced Adenocarcinoma of the Lung
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development of JNJ-64041757 in combination with nivolumab discontinued due to lack of clinical benefit observed in the Phase 1b portion of the study
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108232; 2016-002543-41 (EudraCT Number); 64041757LUC2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Adenocarcinoma of Lung
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + JNJ-64041757 (Experimental): Phase 1b and Phase 2 Group A/Arm 1: Participants will receive separate intravenous (IV) infusions of nivolumab and JNJ-64041757 over approximately 60 minutes during each treatment cycle until disease progression, unacceptable toxicity, protocol violation requiring discontinuation of study treatment, withdrawal of consent, noncompliance with study procedures, or the sponsor terminates the study.
  Interventions: Biological: JNJ-64041757; Drug: Nivolumab
- Nivolumab (Active Comparator): Phase 2 Group B/Arm 2: Participants will receive intravenous (IV) infusions of nivolumab over approximately 60 minutes during each treatment cycle until disease progression, unacceptable toxicity, protocol violation requiring discontinuation of study treatment, withdrawal of consent, noncompliance with study procedures, or the sponsor terminates the study.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Biological: JNJ-64041757 — Participants will receive intravenous (IV) infusions of JNJ-64041757 over approximately 60 minutes during each treatment cycle.
  Other Names: JNJ-757
  Arms: Nivolumab + JNJ-64041757
Drug: Nivolumab — Participants will receive IV infusions of nivolumab over approximately 60 minutes during each treatment cycle.

SUMMARY:
The purpose of this study is to evaluate whether the efficacy of JNJ-757 combined with nivolumab is better than the efficacy of nivolumab monotherapy for participants with mesothelin-positive relapsed/refractory Stage IIIB or Stage IV adenocarcinoma of the lung. The open-label study comprises of two parts i.e. Phase 1b (safety run-in) and Phase 2. Phase1b consists of 1 arm whereas Phase 2 is randomized into 2 groups i.e. Group A and Group B.

DETAILED DESCRIPTION:
This study evaluates safety and efficacy of JNJ-64041757 with nivolumab. The total study duration will be up to 3 years. It will consist of safety run-in and randomized phase which will comprise of Screening phase(Day(D) -28 to D -1),Treatment Phase,End of Adverse Event Evaluation Period (100 D after last dose of nivolumab)and Post-treatment Follow-up Phase(Every 3 Months). The primary hypothesis is that addition of JNJ-640417577 to nivolumab will result in higher objective response rate compared with nivolumab monotherapy in at least one of programmed death receptor ligand 1 subgroups in participants with relapsed or refractory StageIIIB or StageIV adenocarcinoma of lung. The study procedures include blood culture bacterial shedding assessments, pharmacokinetics, immunogenicity, and biomarkers. Safety will be monitored throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Disease-related criteria: Histologically documented adenocarcinoma of the lung; Stage IIIB or Stage IV disease; Biopsy material available for central assessment of programmed death receptor ligand 1 (PD-L1) and mesothelin
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Progressive disease during or after platinum-based doublet chemotherapy
* A woman of childbearing potential must have a negative serum or urine pregnancy test within 14 days before the first dose of nivolumab
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Tumor with activating epidermal growth factor receptor (EGFR) mutation or ALK translocation
* More than 1 prior line of chemotherapy for metastatic disease (Phase 2)
* History of disallowed therapies, as follows: In Phase 1b only: Prior exposure to anti-programmed death receptor-1(PD1), anti programmed death receptor ligand 1 (PD-L1), anti-programmed death receptor ligand 2 (PD-L2), anti-CD137, or anti-cytotoxic T lymphocyte associated antigen 4 (CTLA-4) antibody within 28 days before the first dose of study agent, In Phase 2 only: Prior exposure to anti-PD1, anti PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte associated antigen 4 (CTLA-4) antibody, History of listeriosis or vaccination with a Listeria-based vaccine or prophylactic vaccine within 28 days before the first dose of study agent, Chemotherapy within 28 days before the first dose of study agent, Radiation within 14 days before the first dose of study agent
* History of any other condition that may require the initiation of anti-tumor necrosis factor alpha (TNF alpha) therapies or other immunosuppressant medications during the study
* Active second malignancy within 2 years prior to Cycle 1 Day 1 (Phase 1b) or randomization (Phase 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- United States (3):
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Medical Oncology Associates, PS, Spokane, Washington
- AZ Maria Middelares, Ghent, Belgium
- Spain (6):
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp. Gral. Univ. de Elche, Elche
  - Complejo Hospitalario de Jaen, Jaén
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Son Llatzer, Palma de Mallorca
  - Hosp. Arnau de Vilanova de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial consisted of two parts (Phase 1 b and Phase 2). However, Phase 2 was not conducted due to early termination of the study. All analyses were performed on Phase 1b data.
Groups:
- Phase 1b: JNJ-64041757+ Nivolumab: Participants received nivolumab 240 milligram (mg) intravenous (IV) infusion followed by JNJ-64041757 (1*10^9 colony-forming units [CFUs]) IV infusion on Day 1 and nivolumab 240 mg IV infusion on Day 15 of each 28-day cycle until disease progression, unacceptable toxicity, protocol violation requiring discontinuation of study treatment, withdrawal of consent, noncompliance with study procedures, or the sponsor terminates the study.
Period: Overall Study
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Started | 12
Completed | 0
Not Completed | 12
Not completed — Death | 5
Not completed — Study terminated by sponsor | 3
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  White Non-Hispanic | 11
Region of Enrollment [Count of Participants; unit: Participants]
  SPAIN | 10
  UNITED STATES | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Percentage of Participants With Objective Response
Description: Objective response rate was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST). RECIST for CR - disappearance of all lesions; all lymph nodes were non-pathological in size and normalization of tumor marker level; PR - greater than or equal to (>=) 30 percent (%) decrease in the sum of the diameters of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of nontarget lesions.
Time Frame: Up to 6.8 Months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Percentage of participants | 0

2. Secondary Outcome: Phase 1b: Duration of Objective Response (DOR)
Description: Duration of objective response was defined as the time from initial documentation of a response (CR or PR) to first documented date of disease progression (PD) or death from any cause. RECIST for PD - sum of diameters had increased by >= 20% and >=5 mm from nadir (including baseline if it was smallest sum). Participants with measurable disease: for "unequivocal progression" based on non-target disease, there was an overall level of substantial worsening that merits discontinuation of therapy (if target disease is stable disease [SD]/PR). Participants without measurable disease: for "unequivocal progression" of non-target disease, increase in overall tumor burden must be comparable to increase required for PD of measurable disease. Furthermore, appearance of 1 or more new lesions or unequivocal progression of a non-target lesion.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent. Overall number of participants analyzed is zero, since none of the participants had objective response.
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1b: Number of Participants With Progression-free Survival (PFS) Event (Progressed or Died Before Progression)
Description: Number of participants with PFS event (progressed or died before progression) were reported. PFS - time from date of randomization until date of first documented evidence of PD (or relapse for participants who experience CR during study) or death from any cause, whichever comes first. RECIST for PD - sum of diameters had increased by >= 20% and >=5 mm from nadir (including baseline if it was smallest sum). Participants with measurable disease: for "unequivocal progression" based on non-target disease, there was an overall level of substantial worsening that merits discontinuation of therapy (if target disease is SD/PR). Participants without measurable disease: for "unequivocal progression" of non-target disease, increase in overall tumor burden must be comparable to increase required for PD of measurable disease. Furthermore, appearance of 1 or more new lesions or unequivocal progression of a non-target lesion.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 10

4. Secondary Outcome: Phase 1b: Number of Participants With Overall Survival (OS) Event (Died)
Description: Number of participants with OS event (died) were reported. Overall Survival was defined as the duration from the date of randomization to the date of participant's death due to any cause.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 5

5. Secondary Outcome: Phase 1b: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as adverse events with onset or worsening on or after date of first dose of study treatment.
Time Frame: Up to 6.8 months
Population: Safety analysis set included participants who received at least 1 administration of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 12

6. Secondary Outcome: Phase 1b: Number of Participants With Positive Blood Culture
Description: Number of participants with surveillance cultures positive for listeriosis were reported.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 1

7. Secondary Outcome: Phase 1b: Number of Participants With Bacterial Shedding
Description: Number of participants with bacterial shedding were reported. The shedding of JNJ-64041757 was studied in feces by stool or rectal swab, urine and saliva.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 0

8. Secondary Outcome: Phase 1b: Serum Concentrations of Nivolumab
Description: Nivolumab serum concentrations were reported.
Time Frame: Up to 6.8 months
Population: Pharmacokinetic (PK) population consisted of all participants who received at least 1 dose of study agent and had one PK blood sample available. Although PK samples were collected, but assays were not run due to no longer development of compound.
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 1b: Number of Participants With Anti-nivolumab Antibodies
Description: Number of participants with antibodies to nivolumab were reported.
Time Frame: Up to 6.8 months
Population: The all treated analysis population consisted of participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
Number analyzed (Participants) | 12
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 6.8 months
Description: Safety analysis set included participants who received at least 1 administration of any study medication.
Arm/Group | Phase 1b: JNJ-64041757+ Nivolumab
All-Cause Mortality (participants affected / at risk) | 5/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: JNJ-64041757+ Nivolumab (N=12)
Abdominal Pain (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: JNJ-64041757+ Nivolumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 6
Chills (General disorders) | 7
Fatigue (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 2
Pyrexia (General disorders) | 8
Hepatic Failure (Hepatobiliary disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1
Blood Creatinine Increased (Investigations) | 1
Body Temperature Increased (Investigations) | 1
Weight Decreased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Inferior Vena Caval Occlusion (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Sponsor did not proceed to Randomized phase 2 of study or enroll additional participants in phase 1b as study was stopped early, that resulted in limited evaluation of planned participant-related outcomes, PK, immunogenicity and biomarker analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT03371381/Prot_SAP_000.pdf